CLINICAL TRIAL: NCT04872894
Title: Familial Hypocalciuric Hypercalcemia: Clinical Aspects and Evolution
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-HCF-2020-89
Record Dates: First submitted 2021-03-15; First posted 2021-05-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2021-04

CONDITIONS: Familial Hypocalciuric Hypercalcemia
Keywords: hypercalcemia; Familial Benign Hypercalcemia; Familial hypocalciuric hypercalcemia
MeSH Terms: conditions — Hypocalciuric hypercalcemia, familial, type 1; Hypercalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study. No intervention is performed — Descriptive study in participants with clinical and biochemical suspicion of FHH. Comparison between genotype-negative and genotype-positive participants with clinical and biochemical suspicion of FHH.

SUMMARY:
Familial hypocalciuric hypercalcemia (FHH) is a rare disease (ORPHA#405, www.orpha.net) and most likely underdiagnosed, that clinicians should be aware of in the differential diagnosis of a hypercalcemia. Appropriate identification of the FHH has implications in treatment and also for the family, since it is an automosal-dominant disease, due to mostly a heterozygous loss-of-function mutation of the CASR (calcium-sensing receptor) gene, but also much less freqüent mutations of another two genes (AP2S1 and GNA11). In case of clinical and biochemical suspicion of FHH, a genetic evaluation is mandatory. Nevertheless, an important number of patients, the genetic study is negative. This observational study is intended to perform a descriptive review of cases with clinical and biochemical suspicion of FHH who underwent a genetic study in the usual clinical practice. Clinical, biochemical and radiological characteristics, treatment, follow-up and comorbidities of genotype-negative participants will be compared with genotype-positive cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and biochemical suspicion of FHH who, at the discretion of the physician in routine clinical practice, were asked to perform a genetic evaluation of FHH and whose genetic results are available.

Exclusion Criteria:

* Genetic study of FHH is not available or was not performed despite clinical and biochemical suspicion of FHH.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants with biochemical and clinical suspicion of FHH, namely hypercalcemia, hypophospatemia, normal or elevated parathormone levels and very low urine calcium excretion defined as a calcium creatinine clearance ratio <0.01, and who were asked at discretion of the clinician for a genetic evaluation of any of the FHH causing genes.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Age (years) | 1 year
  Clinical characteristics of genotype-negative and genotype-positive participants with biochemical suspicion of FHH
Gender distribution (%) | 1 year
  Of genotype-negative and genotype-positive participants with biochemical suspicion of FHH
Calcium levels (mg/dL) | Through study completion, an average of 1 year
  Biochemical characteristics. Of genotype-negative and genotype-positive participants with biochemical suspicion of FHH
Parathyroid Ultrasound results | 1 year
  Of genotype-negative and genotype-positive participants with biochemical suspicion of FHH

SECONDARY OUTCOMES:
Treatment modalities used | 1 year
  Of genotype-negative and genotype-positive participants with biochemical suspicion of FHH
FHH associated comorbidities | Through study completion, an average of 1 year
  Of genotype-negative and genotype-positive participants with biochemical suspicion of FHH

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No